CLINICAL TRIAL: NCT02550262
Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor: A Sequential Allocation Trial to Determine the Optimum Interval Time Between Boluses of a Fixed Volume of 10 ml of Bupivacaine 0.0625% Plus Fentanyl 2 mcg/ml.
Brief Title: Programmed Intermittent Epidural Bolus for Labor Analgesia During First Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-01
Record Dates: First submitted 2015-09-02; First posted 2015-09-15 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Labor Pain
Keywords: Epidural; Labor analgesia; Programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine; Fentanyl; Infusion Pumps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 60 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 60-minute interval. The bolus will consist of 10mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump
- 50 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 50-minute interval. The bolus will consist of 10mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump
- 40 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 40-minute interval. The bolus will consist of 10mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump
- 30 minutes (Experimental): The infusion pump will deliver programmed intermittent epidural boluses at a 30-minute interval. The bolus will consist of 10mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml. A PCEA bolus of 5mL of 0.0625% Bupivacaine plus fentanyl 2mcg/ml will also be available.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Device: Infusion pump

INTERVENTIONS:
Drug: Bupivacaine — 0.0625% Bupivacaine plus fentanyl 2mcg/ml
  Other Names: Marcaine
Drug: Fentanyl — 0.0625% Bupivacaine plus fentanyl 2mcg/ml
Device: Infusion pump — Infusion pump set to deliver programmed intermittent epidural boluses (PIEB) plus patient-controlled epidural analgesia (PCEA).
  Other Names: CADD-Solis Ambulatory Infusion Pump

SUMMARY:
Until recently, at Mount Sinai Hospital, epidural analgesia for labor pain was delivered with a pump that could only provide continuous infusion of the freezing medication in combination of pushes of medication activated by the patient, a technique called patient controlled epidural analgesia (PCEA). In the last decade or so, the literature has suggested that this continuous infusion of medication is not as effective as previously thought, and suggested that instead of continuous infusion, intermittent programmed pushes should be used. The investigators now have devices that are able to do that. Programmed intermittent epidural bolus (PIEB) is a new technological advance based on the concept that boluses of freezing medication in the epidural space are superior to continuous epidural infusion (CEI). The new pumps are able to deliver bolus of medication at regular intervals (PIEB), in addition to what the patient can deliver herself (PCEA). Studies have shown that delivering analgesia in this manner can prolong the duration of analgesia, diminish motor block, lower the incidence of breakthrough pain, improve maternal satisfaction and decrease local anesthetic consumption. Based on the information already available in the literature, this study aims to determine the best regimen of PIEB achievable with our standard epidural mixture.

The hypothesis of this study is that there is an optimal interval time between PIEB boluses of 30 to 60 minutes at a fixed volume of 10 ml of our standard epidural mixture that will provide women the necessary drug requirements, thus avoiding breakthrough pain and need for PCEA or physician intervention.

DETAILED DESCRIPTION:
All studies involving PIEB to date have provided an analgesic regimen that delivered an amount of local anesthetic that was below the patient's requirement per hour, as the studies were done in the context of an association with PCEA (Patient controlled epidural anesthesia) as a rescue technique. As a result, PCEA requests were frequent and therefore these studies have not been able to truly understand the pharmacology of the bolus technique in the PIEB regimen, as the PCEA utilized by patients added an extra component to the regimen.

The ideal volume and interval time between PIEB bolus has not yet been established in the literature. Most likely the ideal volume and interval time between PIEB bolus will be specific for each epidural mixture.

At Mount Sinai Hospital, PIEB devices have been recently introduced. Currently our standard epidural mixture is bupivacaine 0.0625% with fentanyl 2mcg/ml. Our current epidural regimen consists of 10 ml continuous infusion per hour, with PCEA boluses of 5 ml and a lock out interval of 10 minutes, for a maximum of 20 ml of the epidural mixture per hour. In this study, the investigators will offer patients 10mL PIEBs of bupivacaine 0.0625% with fentanyl 2mcg/ml at 4 different intervals. PCEA bolus of 5mL of the same solution will also be available. The goal is to establish the ideal PIEB regimen that will be effective for our patient population with our standard epidural mixture.

Finding the best way of using the new device that will be able to provide analgesia for 90% of the parturients will represent a great improvement in labor analgesia. Moreover, there are expectations of having fewer side effects since the PIEB is more effective than CEI.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Full term (≥ 37 weeks gestation)
* nulliparous
* Singleton pregnancy, vertex presentation
* Regular painful contractions occurring at least every 5 minutes
* VAS Pain score at requesting analgesia > 5 (VNPS 0-10)
* Cervical dilatation < 5 cm

Exclusion Criteria:

* Refusal to provide written informed consent.
* Any contraindication to epidural anesthesia
* Accidental dural puncture
* Allergy or hypersensitivity to bupivacaine or fentanyl
* Use of opioids or sedatives within the last 4 hours.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
No request for supplemental analgesia | 6 hours
  No request for supplemental analgesia (PCEA bolus or clinician administered bolus) until the completion of the first stage of labor or until 6 hours following initiation of the programmed intermittent epidural bolus (PIEB).

SECONDARY OUTCOMES:
Sensory block level | 6 hours
  Sensory block to ice will be assessed bilaterally at the mid axillary lines, and the level of block will be the level at which the patient still does not feel cold sensation as compared to a control site (frontal part of the head)
Motor block level assessed using Bromage score | 6 hours
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle.
Hypotension | 6 hours
  A decrease in systolic blood pressure greater than 20% from baseline (defined as an average of 3 readings prior to epidural).
Pain score | 6 hours
  Pain score measured hourly using VNRS (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No